CLINICAL TRIAL: NCT06352918
Title: The Effect of Palmar Grasp Reflex Stimulation on Pain and Comfort Level in Peripherally Inducted Central Catheter (PICC) Care in Preterm Babies
Brief Title: Peripheral Central Catheter (PICC) Care
Acronym: PICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Türkan Kadiroğlu, Principal Investıgator, Ataturk University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/395
Record Dates: First submitted 2024-04-03; First posted 2024-04-08 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: NEWBORN; Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reflex Stimulation (Experimental): Along with the NICU PICC care application procedures, palmar grasp reflex stimulation was performed on all babies by the same researcher, starting one minute before the procedure.
  Interventions: Other: Palmar grasp reflex stimulation
- PICC Care (No Intervention): Without any intervention to the control group, the necessary data were recorded in accordance with the NICU's PICC care application procedures.

INTERVENTIONS:
Other: Palmar grasp reflex stimulation — This initiative is stimulated by applying gentle pressure to the palm of the baby's palm while he or she is awake, lying on a flat surface in a symmetrical supine position.
  Arms: Reflex Stimulation

SUMMARY:
Peripheral Central Catheter (PICC) is one of the painful interventions that are routinely performed repeatedly to establish a safe venous access in preterm babies.Nurses should reduce the pain of babies and ensure their comfort during interventions arising from the necessity of care processes.

Today, it is accepted that tactile stimuli, which have a pain-reducing effect on babies, should be used as a complementary treatment and care method. Palmar grasp reflex is one of the important tactile stimuli to reduce pain and provide comfort in babies. This research will be conducted to examine the effect of palmar grasp reflex stimulation on pain and comfort levels in PICC care in preterm babies.

ELIGIBILITY:
Inclusion Criteria:

* Without congenital defects,
* Not receiving sedation at least 3 hours before PICC care,
* No unexplained crying,
* Without neurological problems,
* Not undergoing surgical intervention,
* Babies with PICC insertion

Exclusion Criteria:

* Having had a painful procedure (invasive procedure, etc.) within the last hour,
* Babies for whom permission was not obtained from the parent through an informed voluntary consent form

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Pain level | 8 months
  Premature Infant Pain Scale-Revision (PIPP-R): It is defined as the gestational age of preterm babies, change in heart rate, change in SPO2 level, initial behavioral state, frowning, squeezing eyes, nasolabial groove.

SECONDARY OUTCOMES:
Comfort | 8 months
  COMFORT neo: Consists of 7 sections: alertness, calmness/agitation, respiratory status, physical movements, muscle tone, facial expression and average heart rate. Each section has 5 items with 1 to 5 points. The cut-off point is 17 points on the comfort scale, with a minimum of 7 and a maximum of 35.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No